CLINICAL TRIAL: NCT00096187
Title: A Phase II Trial of Pemetrexed (ALIMTA®, LY231514, IND #40061) as Salvage Therapy for Failed Low Risk Gestational Trophoblastic Tumor
Brief Title: Pemetrexed Disodium in Treating Patients With Recurrent or Persistent Low-Risk Gestational Trophoblastic Tumor After a Molar Pregnancy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000390347; GOG-0217; GOG-UC0205; LILLY-H3E-US-JMGR
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Gestational Trophoblastic Tumor
Keywords: low risk metastatic gestational trophoblastic tumor; recurrent gestational trophoblastic tumor; nonmetastatic gestational trophoblastic tumor
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — Pemetrexed

INTERVENTIONS:
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well pemetrexed disodium works in treating patients with recurrent or persistent low-risk gestational trophoblastic tumor after a molar pregnancy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of pemetrexed disodium as salvage therapy in patients with persistent or recurrent low-risk post-molar gestational trophoblastic tumor that failed prior dactinomycin or methotrexate.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of unacceptable toxicity or disease progression or until tumor marker levels (human chorionic gonadotropin [hCG]) become normal. Patients receive 2 additional courses beyond the attainment of a normal hCG.

Beginning 7 days before and continuing until 3 weeks after the last dose of pemetrexed disodium, patients also receive oral folic acid daily and cyanocobalamin (vitamin B_12) intramuscularly every 9 weeks.

Patients are followed every 2 weeks for 2 months and then monthly for 10 months.

PROJECTED ACCRUAL: Approximately 17-55 patients will be accrued for this study within 20-50 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of low-risk post-molar gestational trophoblastic tumor, defined as 1 of the following:

  * Increasing human chorionic gonadotropin (hCG) levels on ≥ 3 consecutive measurements taken over ≥ a 2-week period
  * Less than 10% decrease of hCG levels on 4 measurements taken over ≥ a 3-week period
* Persistent or recurrent disease
* Histologically confirmed complete or partial mole on initial evacuation

  * Prior pregnancy ≤ 12 months ago
* No histologically confirmed choriocarcinoma or placental site trophoblastic tumor on initial evacuation
* Failed only 1 prior dactinomycin or methotrexate therapy (with or without leucovorin calcium)
* WHO score 2-6
* No evidence of metastatic disease, except to the lung or vagina, on physical exam, chemistry, chest X-ray, and ultrasound

  * No liver, spleen, brain, kidney, or gastrointestinal tract metastases
  * No more than 8 metastatic lesions

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* GOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Granulocyte count ≥ 1,500/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN

Renal

* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 45 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* No significant infection
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic filgrastim (G-CSF) unless for recurrent neutropenic complications
* No concurrent prophylactic thrombopoietic agents unless for recurrent grade 4 thrombocytopenia

Chemotherapy

* See Disease Characteristics
* At least 7 days since prior dactinomycin or methotrexate (with or without leucovorin calcium) and recovered
* No prior pemetrexed disodium
* No other prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 14 days since prior radiotherapy and recovered
* No prior radiotherapy to ≥ 25% of the bone marrow

Surgery

* Recovered from prior surgery

Other

* No nonsteroidal anti-inflammatory drugs or salicylates for 2 days (or 5 days for drugs with a long half-life) before, during, and for 2 days after pemetrexed disodium administration

  * Concurrent low-dose aspirin (≤ 325 mg/day) allowed

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-07-23 (Actual)

PRIMARY OUTCOMES:
Activity
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center; Allan Covens, MD — Toronto Sunnybrook Regional Cancer Centre
Locations (25):
- United States (25):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas